CLINICAL TRIAL: NCT00631527
Title: Sunitinib, Hormonal Ablation and External Beam Radiation Therapy for High-Risk and Locally Advanced Prostate Cancer
Brief Title: Sunitinib Malate, Hormone Ablation and Radiation Therapy in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0684; NCI-2010-01524 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radiation Therapy; RT; Radiotherapy; Hormone Ablation; Sunitinib Malate; Leuprolide; Lupron; Zoladex; Goserelin; Casodex; Bicalutamide; SU011248; Sutent; Angiogenesis inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Goserelin; Sunitinib; bicalutamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib Malate, Hormone Ablation + RT (Experimental): Sunitinib Malate + Hormone Ablation (Leuprolide or Goserelin + Bicalutamide) + Radiation Therapy (RT)
  Interventions: Drug: Leuprolide; Drug: Goserelin; Drug: Sunitinib Malate; Drug: Casodex; Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Leuprolide — Injections given through a needle in the muscle every 3 months.
  Other Names: Lupron
Drug: Goserelin — Subcutaneous injections given once every 3 months.
  Other Names: Zoladex
Drug: Sunitinib Malate — Starting dose of 12.5 mg by mouth daily for 4 weeks
  Other Names: SU011248; Sutent
Drug: Casodex — Once a day by mouth for 2 weeks.
  Other Names: Bicalutamide
Radiation: Radiation Therapy (RT) — Radiation treatment once daily over a period of 8 weeks.
  Other Names: Radiotherapy

SUMMARY:
The goal of this clinical research study is to learn the safety of adding 3 different dose-levels of Sutent® (sunitinib malate) to a combination of hormone therapy and radiation in patients with prostate cancer.

DETAILED DESCRIPTION:
The Study Drugs:

Sunitinib malate is designed to block pathways that control important events such as the growth of blood vessels that are essential for the growth of cancer.

Luteinizing Hormone-Releasing Hormone (LHRH) Analogues like Lupron® (leuprolide) and Zoladex® (goserelin) are hormonal treatments used to help stop the body from making testosterone (male sex hormones) in the body. Prostate cancer cells need testosterone to survive.

Anti-Androgen drugs, like Casodex® (bicalutamide) also stop cell growth by blocking male hormones like testosterone.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will be assigned to a study group. The group you are assigned to and dose of sunitinib malate you receive will depend on when you join this study. Three (3) dose levels of sunitinib malate will be tested. The first group of participants will receive the lowest dose of sunitinib malate. The next group enrolled will receive a higher dose of sunitinib malate, if no intolerable side effects were seen.

Before you begin taking sunitinib, you will begin receiving hormone therapy. You will receive leuprolide or goserelin. Leuprolide is given through a needle in your muscle, and goserelin is given through a needle under the skin in the abdomen. You will receive 1 of these injections every 3 months. Which hormonal drug you are given (leuprolide or goserelin) will be assigned by your doctor and/or will depend on your insurance coverage.

You may also receive bicalutamide. This will be left up to the doctor. You will take bicalutamide by mouth once a day for 2 weeks (with or without food).

After at least 4 weeks of hormone therapy have been given, you will begin taking sunitinib malate in combination with the hormone therapy. You will take sunitinib malate once a day (either with or without food) for 16 weeks in a row.

Radiation Therapy:

After 4 weeks of combined treatment with sunitinib and hormone therapy, you will begin radiation treatments. Radiation treatments will be given once a day, 5 days a week, for about 8 weeks. Each treatment will take 20-30 minutes. This procedure will be discussed with you in more detail. You will continue taking sunitinib and hormone therapy while you are on radiation treatments.

Study Visits:

On the day you start treatment with sunitinib, you will have the following tests and procedures performed:

* You will have a physical exam, including measurements of your blood pressure and weight.
* You will be asked about any side effects you may have had since your last visit.
* Blood (about 1 teaspoon) will be drawn for routine tests.

About Day 15 of treatment with sunitinib, and on the day you begin radiation therapy (before your first treatment), you will have the following tests and procedures performed:

* You will have a physical exam, including measurements of your blood pressure and weight.
* You will be asked about any side effects you may have had since your last visit.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Every 2 weeks during radiation therapy, you will have the following tests and procedures performed:

* You will have a physical exam, including measurements of your blood pressure and weight (every 2 weeks)
* You will have blood drawn (about 2 teaspoons) for routine testing.
* You will be asked about any side effects you may have had since your last visit.

About 4 weeks after you stop radiation therapy, you will have the following test and procedures performed:

* You will have a physical exam, including measurements of your blood pressure and weight.
* Blood (about 2 teaspoons) and urine will be collected for routine tests. The blood testing will include measurement of prostatic specific antigen (PSA) and testosterone levels.
* You will be asked about any side effects you have had since your last visit.

Length of Study:

You will continue taking sunitinib malate on this study for a total of 16 weeks. Radiation treatments will last for up to 8 weeks. Hormone injections will continue for a period of 2 years. You will be taken off this study if intolerable side effects occur or the disease gets worse.

Long-Term Follow-up:

You will be followed every 6 months via telephone call and/or a review of your medical record. If contacted, you will be asked about any side effects you have had, or therapies you may have had since stopping treatment on this study. You will be followed for up to 10 years once you have taken sunitinib malate for 20 weeks.

This is an investigational study. Sunitinib malate is FDA approved and commercially available for the treatment of adults with kidney cancer.

Bicalutamide, leuprolide, and goserelin are FDA approved and commercially available for use in prostate cancer.

Up to 22 patients will be enrolled in this multicenter trial. Up to 12 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate with the following high-risk features are eligible: clinical T2c, clinical or pathological T3 or T4 disease OR Gleason 8-10 disease OR PSA > 20ng/ml.
2. Patients must have no evidence of metastatic disease by clinical and radiological staging including Chest X-ray, Bone scan and CT Scan of the Abdomen and Pelvis.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
4. Calculated Creatinine clearance > 35cc/min, Absolute neutrophil count > 1,500/mm^3, Platelets >/= 100,000/mm^3, AST/ALT < 2.5 x upper normal limit (UNL), Total bilirubin within normal limits (WNL).
5. No standard contraindications to radiation therapy including prior radiation therapy, inflammatory bowel disease, irritable bowel syndrome, or and collagen vascular disease.
6. Patients must be at least 18 years of age
7. Patients may have had up to 8 weeks of hormonal therapy defined as luteinizing-hormone releasing hormone or other medical castration therapy prior to registration.

Exclusion Criteria:

1. Prior VEGFR/PDGFR inhibitor or other investigational therapy.
2. Inability to take oral medication
3. Chronically uncontrolled hypertension, defined conventionally as consistent/repeated systolic pressures above 140 mmHg or diastolic pressures above 90 mmHg despite anti-hypertensive therapy. This may be established with home BP readings. There is no criterion related to a specific BP result required for eligibility, nor are acute BP elevations that are related to iatrogenic causes, acute pain, or other transient reversible causes considered an exclusion criteria. The intent is to exclude patients with chronically uncontrolled hypertension that might be further exacerbated by Sunitinib.
4. Left Ventricular Ejection Fraction </= 40%, symptomatic congestive heart failure or symptomatic ischemic heart disease, deep venous thrombosis or pulmonary embolism in the last 12 months.
5. Known human immunodeficiency virus infection, alcoholism, chronic active hepatitis or liver cirrhosis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as defined by Dose Limiting Toxicity (DLT) | 8 weeks
  DLT defined as inability to complete the schedule course of radiation therapy for toxicity of any grade. If < 2 patients in initial cohort of 6 experience DLT then a subsequent dose-level cohort initiated. If 2 or more patients in a cohort experience DLT then further accrual to that cohort curtailed and no higher dose level examined. Maximum tolerated dose (MTD) for oral sunitinib in combination with radiation and hormone ablation defined as highest dose level in which 6 patients have been treated with 2 or less than 2 instances of DLT.
  DLT for the purposes of dose-escalation or calculation of the maximum tolerated dose (MTD) defined as any medically unmanageable Grade 2 toxicity or any Grade 3 or 4 toxicity experienced during the 8 week period of combined hormone ablation, Sunitinib, and radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Karlou M, Tzelepi V, Efstathiou E. Therapeutic targeting of the prostate cancer microenvironment. Nat Rev Urol. 2010 Sep;7(9):494-509. doi: 10.1038/nrurol.2010.134. PMID 20818327
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org